CLINICAL TRIAL: NCT05466422
Title: A Multiple Ascending Dose Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-2214 in Adults With Mild Cognitive Impairment or Mild-to-Moderate Alzheimer's Disease
Brief Title: A Study of MK-2214 in Adults With Mild Cognitive Impairment or Mild-to-Moderate Alzheimer's Disease (MK-2214-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2214-002; MK-2214-002 (Other: MSD)
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-2214 (Experimental): Participants will receive MK-2214 administered in escalating doses as an intravenous (IV) infusion on Days 1, 29, and 57.
  Interventions: Biological: MK-2214
- Placebo (Placebo Comparator): Participants will receive placebo as an IV infusion on Days 1, 29, and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MK-2214 — MK-2214 in escalating doses as an IV infusion on Days 1, 29, and 57
  Arms: MK-2214
Drug: Placebo — Placebo as an IV infusion on Days 1, 29, and 57
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of MK-2214 in adults with mild cognitive impairment (MCI) or mild-to-moderate Alzheimer's Disease (AD). The primary hypothesis (Part 1) is that at a generally well tolerated dose level, the true geometric mean concentration at Day 85 of MK-2214 in cerebrospinal fluid is >0.3 nanomolar (nM).

ELIGIBILITY:
Inclusion Criteria:

* Participant is in overall good health based on medical history and laboratory safety tests
* BMI between 18.5 and 35 kg/m^2

Part 1 (MCI and Mild to Moderate AD) Only:

* History of cognitive and functional decline with gradual onset and slow progression for at least one year before Screening
* Have an Mini-Mental State Examination (MMSE) >12 at the prestudy visit
* Modified Hachinski Ischemic Score (MHIS) score <4 at the prestudy visit

Exclusion Criteria:

* Based on clinical interview and Columbia-Suicide Severity Rating Scale (C-SSRS), has reported suicidal ideation with intent, with or without a plan or method
* History of unstable or poorly controlled endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, renal, respiratory, or genitourinary abnormalities or diseases
* History of clinically significant active neurological disease (except for AD or MCI for participants in Part 1)
* History of clinically significant active autoimmune disease requiring ongoing systemic immunosuppressant therapy
* History of cancer (malignancy)
* History of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Positive test(s) for Hepatitis B Surface Antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy visit
* Has a contraindication to lumbar dural puncture, such as coagulopathy, concomitant anticoagulation beyond low dose aspirin, thrombocytopenia, or other factors that could preclude safe lumbar puncture
* Currently receiving or has received aducanumab or another anti-amyloid therapy within the last 6 months
* Has a history of receiving biological therapy within 3 months or 5 half-lives (whichever is longer) or any human immunoglobulin preparation within the last year
* Has received any non-live vaccine starting from 14 days prior to first study intervention or is scheduled to receive any non-live vaccine through 14 days following the final dose of study intervention. Exception: COVID-19 and influenza vaccines may be administered
* Is receiving systemic immunosuppression, including corticosteroids exceeding physiologic replacement doses

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience At Least One Adverse Event (AE) | Up to approximately 297 days
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 57 days
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Serum Area Under the Concentration-Time Curve of MK-2214 from Time 0 to 28 Hours (AUC0-28) After First and Third Dose | At designated time points (up to 85 days)
  AUC is a measure of the extrapolated mean concentration in serum. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine AUC0-28 of MK-2214.
Serum Maximum Concentration (Cmax) of MK-2214 After First and Third Dose | At designated time points (up to 85 days)
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine Cmax of MK-2214.
Serum Time to Maximum Concentration (Tmax) of MK-2214 After First and Third Dose | At designated time points (up to 85 days)
  Tmax is the amount of time required to reach Cmax. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine Tmax of MK-2214.
Serum Apparent Terminal Half-Life (t1/2) of MK-2214 After First and Third Dose | At designated time points (up to 85 days)
  t1/2 is the time required for 50% of drug to be cleared from serum. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine t1/2 of MK-2214.
Concentration of MK-2214 in Cerebrospinal Fluid (CSF) at Day 85 (C85d) | Day 85
  CSF concentration of MK-2214 will be presented for Day 85.
Percentage change from baseline to Day 29 in free phospho-tau in CSF | Baseline and Day 29 pre-dose
  Free phospho-tau in CSF will be determined for participants using the individual percent of baseline values (100* free phospho-tau / baseline).
Percentage change from baseline to Day 85 in free phospho-tau in CSF | Baseline and Day 85
  Free phospho-tau in CSF will be determined for participants using the individual percent of baseline values (100* free phospho-tau / baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (12):
- United States (12):
  - California Clinical Trials Medical Group managed by PAREXEL-PAREXEL International ( Site 0007), Glendale, California
  - Collaborative Neuroscience Research, LLC ( Site 0009), Los Alamitos, California
  - NRC Research Institute ( Site 0015), Orange, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0001), Hallandale, Florida
  - Research Centers of America ( Hollywood ) ( Site 0004), Hollywood, Florida
  - K2 Medical Research ( Site 0005), Maitland, Florida
  - Charter Research - Winter Park ( Site 0012), Orlando, Florida
  - Progressive Medical Research-Alzheimer's Team ( Site 0013), Port Orange, Florida
  - Charter Research - Lady Lake ( Site 0011), The Villages, Florida
  - CenExel iResearch, LLC ( Site 0002), Decatur, Georgia
  - Global Medical Institutes LLC; Princeton Medical Institute ( Site 0003), Princeton, New Jersey
  - Neuro-Behavioral Clinical Research ( Site 0016), North Canton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/